CLINICAL TRIAL: NCT02683395
Title: A Phase 1b/2a, Two-Part, Dose Escalation and Expansion Study to Assess the Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of PLX51107 in Subjects With Advanced Hematological Malignancies and Solid Tumors
Brief Title: A Study of PLX51107 in Advanced Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Plexxikon (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PLX122-01
Record Dates: First submitted 2016-02-12; First posted 2016-02-17 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Solid Tumors; Acute Myeloid Leukemia; Myelodysplastic Syndrome; Non-Hodgkin's Lymphoma
Keywords: PLX51107; Acute Myeloid Leukemia; Myelodysplastic Syndrome; Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin | interventions — PLX51107

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group A (Experimental): Open label, sequential PLX51107 dose escalation in approximately 30 solid tumor subjects.
  Interventions: Drug: PLX51107
- Treatment Group B (Experimental): Open label, sequential PLX51107 dose escalation in approximately 30 subjects with acute myeloid leukemia (AML) or high-risk myelodysplastic syndrome (MDS).
  Interventions: Drug: PLX51107

INTERVENTIONS:
Drug: PLX51107

SUMMARY:
The purpose of this research study is to evaluate safety, pharmacokinetics, pharmacodynamics, and preliminary efficacy of the investigational drug PLX51107 in subjects with advanced solid tumors (including lymphoma), and advanced hematological malignancies

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of a relapsed or refractory malignancy in 1 of 2 treatment groups:

   1. Group A: Subjects with any solid tumor (including lymphomas).
   2. Group B: Subjects with relapsed or refractory AML, Subjects with relapsed or refractory high-risk MDS, defined as revised International Prognostic Scoring System (IPSS-R) intermediate or greater disease.
2. Age ≥18 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
4. Life expectancy ≥3 months in the judgment of the investigator.
5. Adequate organ function.
6. Group A subjects must have measurable or evaluable disease per the appropriate disease criteria.
7. Women of child-bearing potential must have a negative serum pregnancy test at Screening and must agree to use an effective form of contraception from the time of the negative pregnancy test up to 6 months after the last dose of study drug. Effective forms of contraception include abstinence, hormonal contraceptive in conjunction with a barrier method, or a double barrier method. Women of non-child-bearing potential may be included if they are either surgically sterile or have been postmenopausal for ≥1 year.
8. Fertile men must agree to use an effective method of birth control during the study and for up to 6 months after the last dose of study drug.
9. All associated clinically significant toxicity from previous cancer therapy must be resolved (to ≤Grade 1 or baseline) prior to study treatment administration (Grade 2 alopecia is allowed).
10. Willingness and ability to provide written informed consent prior to any study-related procedures and to comply with all study requirements.

Exclusion Criteria:

1. Prior exposure to a bromodomain inhibitor, such as OTX-015 or CPI-0610.
2. Allogenic or autologous transplant for hematological malignancy with infusion of stem cells within 90 days before Cycle 1 Day 1, or on active immunosuppressive therapy for graft-versus-host disease (GVHD) or GVHD prophylaxis within 2 weeks of Cycle 1 Day 1.
3. Known uncontrolled fungal, bacterial, and/or viral infection ≥Grade 2.
4. Uncontrolled autoimmune hemolytic anemia or thrombocytopenia.
5. For Group A: Subjects with a history of brain metastases are ineligible. This includes previously treated brain metastases. For Group B (subjects with AML): Active symptomatic CNS involvement of AML. Subjects with previously treated leptomeningeal disease that has been effectively treated are eligible.
6. A diagnosis of acute promyelocytic leukemia (APL) or chronic myeloid leukemia (CML) in blast crisis.
7. Known or suspected allergy to the investigational agent or any agent given in association with this trial.
8. Women who are pregnant or are breast feeding.
9. Clinically significant cardiac disease
10. Inability to take oral medication or significant nausea and vomiting, malabsorption, or significant small bowel resection that, in the opinion of the Investigator, would preclude adequate absorption.
11. Subject with known human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) infection or is known to be a carrier of hepatitis B or C.
12. Strong CYP3A4 and CYP2C8 inhibitors or inducers or CYP3A4 substrate drugs with a narrow therapeutic range taken within 14 days or 5 drug half-lives before start of study drug.
13. Active secondary malignancy
14. Major surgery or significant traumatic injury within 14 days prior to therapy
15. Receipt of anti-cancer therapy 14 days prior to Cycle 1 Day 1
16. Presence of any other medical, psychological, familial, sociological, or geographic condition potentially hampering compliance with the study protocol Subjects who are participating in any other therapeutic clinical study (observational or registry trials are allowed).
17. Subjects who have Burkitt's lymphoma or Burkitt-like lymphoma.
18. Subjects on active anticoagulation therapy including warfarin, factor Xa inhibitors, thrombin inhibitors, or heparin.
19. Subjects with documented hepatic metastases involving >50% of the hepatic parenchyma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-03; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Safety of PLX51107 as measured by adverse events and serious adverse events. | 1 year
Area under the concentration-time curve (AUC) of PLX51107. | 1 year
Maximum observed concentration (Cmax) of PLX51107. | 1 year
Time to peak concentration (Tmax) of PLX51107. | 1 year
Half life (t1/2) of PLX51107. | 1 year

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 1 year
  ORR is defined as the total number of patients with the best overall response according to standard criteria for the relevant malignancy divided by the total number of treated patients and expressed as a percentage.
Duration Of Response (DOR). | 1 year
  DOR is defined as the time from the initial objective response to disease progression or death, whichever occurs first.
Progression-Free Survival (PFS). | 1 year
  PFS time is defined as the time from the first dose of PLX51107 to disease progression or death, whichever occurs first.
Overall Survival (OS). | 1 year
  OS is defined as the first dose of study drug until the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Columbia University Medical Center, New York, New York
  - The Ohio State University Stephanie Spielman Comprehensive Breast Center, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - MUSC/ Hollings Cancer Center, Charleston, South Carolina
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided